CLINICAL TRIAL: NCT03263689
Title: The Analgesic Effects of Intrathecal Morphine in Comparison to Ultrasound-guided Transversus Abdominis Plane Block After Cesarean Section: a Randomized Controlled Trial at a Ugandan Regional Referral Hospital
Brief Title: Transversus Abdominis Plane Block Versus Spinal Morphine After Caesarean Section : A Comparison Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mbarara University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MUST/19/08-14
Record Dates: First submitted 2017-08-16; First posted 2017-08-28 (Actual); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Pregnancy, Ceasarian Section, Anaesthesia
MeSH Terms: interventions — Injections, Spinal

STUDY DESIGN:
Intervention Model Description: The patients in the intrathecal morphine (ITM group) were given a sham block, while the patients in the TAP group were given a TAP block. Sham blocks consisted of a non-invasive ultrasound scan. A blunt needle was gently pressed on either side of the abdomen. Bilateral TAP blocks were placed after ultrasound location of the transversus abdominis and internal oblique muscles, with the injection sites in the Triangle of Petit located at the lateral edge of the mid-abdomen. Following negative aspiration for blood, the local anaesthetic (0.25% bupivacaine with 1:200000 epinephrine) was injected in the transversus abdominis plane under ultrasound visualization in 5 cc aliquots for a total volume of 15cc per side.
Who Masked: Participant
Masking Description: The subjects were randomly assigned to a study group (intrathecal morphine - ITM group - or TAP - TAP group) by a computer random number generator. Patients were blinded to their study allocation. Those in the ITM group were given 100 micrograms of preservative-free morphine in addition to the local anaesthesia (plain hyperbaric bupivacaine 10mgs) intrathecally during the spinal anaesthesia. The TAP group were given only local anaesthesia (plain hyperbaric bupivacaine 10 mgs) during the spinal anaesthesia.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intervention (Experimental): ITM group were given
  1. Local anaesthesia (plain hyperbaric bupivacaine 10mgs) intrathecally during the spinal anaesthesia
  2. 100 micrograms of preservative-free morphine.
  Interventions: Drug: Intrathecal morphine
- Control (Active Comparator): TAP group were given only local anaesthesia (plain hyperbaric bupivacaine 10 mgs) during the spinal anaesthesia.
  Interventions: Drug: Intrathecal morphine

INTERVENTIONS:
Drug: Intrathecal morphine — ITM group were given 100 micrograms of preservative-free morphine in addition to the local anaesthesia (plain hyperbaric bupivacaine 10mgs) intrathecally during the spinal anaesthesia
  Other Names: Intrathecal

SUMMARY:
Many counties in sub-Saharan Africa have very limited post-operative nursing capacity, and relatively little data have been published about post-operative maternal pain control in these settings. Cesarean section is the most common type of major operation at our institution, Mbarara Regional Referral Hospital (MRRH), in south-western Uganda.Nursing ward staffing capacity is low, with much basic nursing care provided by families and friends of patients. The investigators conducted a study to examine the impact of ITM versus TAP block in a setting of limited formal nursing oversight.

DETAILED DESCRIPTION:
Intrathecal morphine (ITM), administered as a part of spinal anesthesia for caesarian section, can produce significant post-operative analgesia for several hours. The Tranversus Abdominis Plane (TAP) Block can also provide prolonged post-operative pain control. A small number of published studies comparing analgesic outcomes after cesarian section with ITM or TAP block have reported variable results.Moreover, these studies have been conducted in countries with extensive post-operative nursing care.

Many counties in sub-Saharan Africa have very limited post-operative nursing capacity, and relatively little data have been published about post-operative maternal pain control in these settings. Cesarean section is the most common type of major operation at our institution, Mbarara Regional Referral Hospital (MRRH), in south-western Uganda.Nursing ward staffing capacity is low, with much basic nursing care provided by families and friends of patients. The investigators conducted a study to examine the impact of ITM versus TAP block in a setting of limited formal nursing oversight.

ELIGIBILITY:
Inclusion Criteria:

1. Women between the age of 18-45;
2. Greater than 50 kilograms in weight;
3. Routine spinal anesthetic without sedation for an uncomplicated caesarean delivery via a low, transverse abdominal incision (Pfannenstiel);
4. In good health with no major medical problems including gastric ulcers, liver or renal dysfunction
5. Able to communicate freely with a provided non-family member interpreter fluent in the patient's language so that informed consent may be obtained

Exclusion Criteria:

1. Patients with allergies to bupivacaine, paracetamol, or diclofenac;
2. Patients undergoing a surgical approach is other than a low, transverse abdominal incision (Pfannenstiel);
3. Pre-eclampsia, uterine rupture, placental abruption with this pregnancy;
4. Prior complicated abdominal surgery;
5. Medical history of gastric ulcers, liver or kidney dysfunction; and
6. Patient refusal to be involved in the study. Failure to attain informed consent from the patient due to age or level of consciousness
7. Voluntary or involuntary withdraw from the study
8. Referral to another health centre or Hospital for further management.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant women in labor with indication for ceasarian section
Enrollment: 130 (Actual)
Dates: Start 2014-03-15 (Actual); Primary Completion 2016-06-20 (Actual); Study Completion 2016-06-20 (Actual)

PRIMARY OUTCOMES:
Pain measurement | at 8 hours after intervention
  Pain measurement using the numerical rating scale (NRS).
Pain measurement | at 16 hours after intervention
  Pain measurement using the numerical rating scale (NRS).
Pain measurement | at 24 hours after intervention
  Pain measurement using the numerical rating scale (NRS)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Kwikiriza, MD, Principal Investigator — Mbarara University of Science and Technology

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared after relevant permissions have been obtained